CLINICAL TRIAL: NCT01487265
Title: Phase II Trial of Erlotinib and BKM120 in Patients With Advanced Non Small Cell Lung Cancer Previously Sensitive to Erlotinib
Brief Title: Trial of Erlotinib and BKM120 in Patients With Advanced Non Small Cell Lung Cancer Previously Sensitive to Erlotinib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LUN 214
Record Dates: First submitted 2011-12-01; First posted 2011-12-07 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-02

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Erlotinib; BKM120; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — NVP-BKM120; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BKM120 and Erlotinib (Experimental): Cycle 1: BKM120 80 mg PO daily; Erlotinib 100mg PO daily
  Cycles 2 and beyond: BKM120 100 mg PO daily; Erlotinib 100mg PO daily
  Interventions: Drug: BKM120 and Erlotinib

INTERVENTIONS:
Drug: BKM120 and Erlotinib — BKM120 and Erlotinib will be given once daily. Erlotinib 100 mg PO will be administered. During Cycle 1-Week 1 all patients will receive 80 mg PO daily BKM120. After the first week of Cycle 1, the dose of BKM120 will escalate to 100 mg PO daily and treatment will continue as long as there are no unexpected or prohibitive toxicities, or disease progression.
  Other Names: Buparlisib (BKM 120) and Tarceva (erlotinib)

SUMMARY:
Preclinical data in lung cancer cell lines showed that EGFR mutation can potentially be a positive predictor for sensitivity to BKM120. Furthermore, when the erlotinib-resistant model H1975 (LR858 and T790M mutation) was treated with BKM120, significant tumor control was observed (Novartis internal data). Therefore, combining BKM120 with erlotinib could potentially down-modulate PI3K-Akt activity resulting in a synergistic effect on cell growth inhibition and enhancing the response to erlotinib.

DETAILED DESCRIPTION:
This is a multicentered, open-label, non-randomized Phase II study of BKM120 and erlotinib in patients with advanced NSCLC previously sensitive to erlotinib. After six patients are enrolled and complete one treatment cycle a safety analysis of adverse events (AEs) will be conducted to assure there are no unexpected or prohibitive toxicities of the combination. The planned study enrollment will continue to up to 37 patients. Duration of a patient's participation in the study will vary. Treatment will continue as long as the patient is benefitting from the treatment, has no evidence of disease progression, and does not meet any criteria for discontinuation or withdrawal.

ELIGIBILITY:
Inclusion Criteria:

Patients must have recovered to Grade 1 or better from any adverse events (except alopecia) related to prior antineoplastic therapy before screening procedures are initiated.

1. Patients with progressive NSCLC (any histology)
2. Prior sensitivity to erlotinib or gefitinib or other EGFR TKI. Sensitivity is defined as follows:

   * Patients treated with erlotinib (or gefitinib or other EGFR TKI) for any duration in the presence of a known EGFR activating mutation that confers sensitivity to TKI treatment. These include, but are not limited to mutations in L858R (Exon 21); Exon 19 deletion; G719S, G719A, G719C mutations (Exon 19);or L861Q (laboratory report required at enrollment).
   * Prior treatment with erlotinib (or gefitinib, or other EGFR TKI), regardless of mutation status, where there was ≥6 months of disease control (no disease progression).
3. At least one site of measurable disease as defined by RECIST criteria Version 1.1
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 2
5. Archival tumor tissue available for correlative testing (analysis of resistance mechanism to erlotinib).
6. Failure of at least 1, and no more than 3, prior systemic treatments for advanced disease (either due to progressive disease or toxicity).
7. Male or female ≥18 years of age.
8. Patients may have received radiation for palliation prior to starting study drug if they have recovered from the side effects of such therapy. Time from last palliative radiation to beginning of study treatment should be ≥1 week. Patients may have received prior wide-field radiation prior to starting study drug if they have recovered from the side effects of such therapy. Time from last wide-field radiation to beginning of study treatment should be ≥2 weeks.
9. Fasting plasma glucose (FPG) ≤120 mg/dL (6.7 mmol/L)
10. Adequate hematologic, hepatic and renal function.
11. Total calcium (corrected for serum albumin) WNL (bisphosphonate use for malignant hypercalcemia control is allowed)
12. Magnesium ≥ the lower limit of normal (LLN)
13. Potassium WNL for the institution
14. Serum amylase and lipase ≤ ULN
15. Ability to swallow oral medication
16. Fertile males, defined as all males physiologically capable of conceiving offspring, must use condoms during treatment, and for an additional 24 weeks (6 months in total after study drug discontinuation), and should not father a child in this period.
17. Female patients who are not of child-bearing potential, and female patients of child-bearing potential who agree to use adequate contraceptive measures, who are not breastfeeding, and who have a negative serum or urine pregnancy test performed within 48 hours prior to start of treatment.
18. Willingness and ability to comply with study and follow-up procedures.
19. Ability to understand the investigational nature of this study and give written informed consent.

Exclusion Criteria:

1. Prior treatment with a phosphatidylinositide 3-kinase (PI3K) inhibitor
2. Known hypersensitivity to BKM120, and/or erlotinib/gefitinib
3. Failure to recover to Grade 1 or better from any AEs (except alopecia) related to previous antineoplastic therapy before screening procedures are initiated.
4. Untreated brain metastases. Patients with treated brain metastases may participate in this study, if the patient is ≥2 weeks from therapy completion (including radiation and/or surgery), has recovered from all effects of treatment, is clinically stable at the time of study entry, and is not receiving high-dose steroid therapy (patients on a low stable dose of steroids may be enrolled).
5. Acute or chronic liver or renal disease or pancreatitis
6. The following mood disorders, as judged by the Investigator or a Psychiatrist, or as a result of patient's mood assessment questionnaire:

   * Medically documented history of active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (immediate risk of doing harm to others)
   * ≥ Grade 3 anxiety
   * Meets the cut-off score of ≥10 12 in the Patient Health Questionnaire (PHQ-9) or a cut-off of ≥15 in the Generalized Anxiety Disorder Assessment (GAD-7) mood scale, respectively, or selects a positive response of "1, 2, or 3" to question number 9 regarding potential for suicidal thoughts in the PHQ-9 (independent of the total score of the PHQ-9) will be excluded from the study.
7. Active cardiac disease including any of the following:

   * Angina pectoris that requires the use of anti-anginal medication
   * Ventricular arrhythmias except for benign premature ventricular contractions
   * Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication
   * Conduction abnormality requiring a pacemaker
   * Valvular disease with documented compromise in cardiac function
   * Symptomatic pericarditis
   * Uncontrolled hypertension
8. History of cardiac dysfunction including any of the following:

   * Myocardial infarction within the last 6 months
   * History of documented congestive heart failure (New York Heart Association functional classification III-IV) within the last 6 months
   * Documented cardiomyopathy
   * Stroke or transient ischemic attack within the past 6 months
9. Poorly controlled diabetes mellitus (HbA1c >8%)
10. Currently taking therapeutic doses of warfarin sodium or any other coumadin-derivative anticoagulant. Therapy with low molecular weight heparin (LMWH), rivaroxaban, or fondaparinux is allowed.
11. Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g., active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with the protocol
12. Diarrhea ≥ Grade 2.
13. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drugs (e.g., Crohn's disease, ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
14. Prior treatment with any hematopoietic colony-stimulating growth factors (e.g., G-CSF, GM-CSF) ≤1 week prior to starting study drug. Erythropoietin or darbepoetin therapy, if initiated at least 1 week prior to enrollment, may be continued.
15. Currently receiving treatment with medication with a known risk to prolong the QT interval or inducing Torsades de Pointes and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug.
16. Patients who have taken herbal medications and certain fruits within 7 days prior to starting study drug. Herbal medications include, but are not limited to, St. John's Wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng. Fruits include the CYP3A inhibitors: Seville oranges, grapefruit, pummelos, or exotic citrus fruits.
17. Currently treated with drugs known to be strong inhibitors or inducers of isoenzyme CYP3A, and the treatment cannot be discontinued or switched to a different medication prior to starting study drug. (Concurrent treatment with moderate or weak inhibitors of CYP3A is allowed).
18. Chemotherapy or targeted anticancer therapy ≤4 weeks (6 weeks for nitrosourea, antibodies or mitomycin-C) prior to starting study drug must recover to a Grade 1 before starting the study (with the exception of EGFR targeting TKIs).
19. Patients who have received any continuous or intermittent small molecule therapeutics (excluding monoclonal antibodies or EGFR targeting TKIs) ≤21 days or 5 half-lives (whichever is shorter) prior to starting study drug or who have not recovered from side effects of such therapy. A minimum of 10 days between termination of study drug and administration of BKM120/erlotinib is required.
20. Oral contraception, injected or implanted hormonal methods are not allowed as BKM120 potentially decreases the effectiveness of hormonal contraceptives.
21. Any condition that would prevent patient comprehension of the investigative nature of the study and its associated risks or prevent the ability to comply with study and/or follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-03; Primary Completion 2016-05-31 (Actual); Study Completion 2017-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Spigel, MD, Study Chair — SCRI Development Innovations, LLC
Locations (7):
- United States (7):
  - Florida Cancer Specialists South, Fort Myers, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Florida Cancer Specialists North, St. Petersburg, Florida
  - Florida Cancer Specialists East, West Palm Beach, Florida
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Center for Cancer and Blood Disorders, Fort Worth, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Erlotinib + BKM120: BKM120, administered 80 mg by mouth (PO) daily during the first week of Cycle 1, then escalated to 100 mg PO daily. Erlotinib, administered 100 mg PO daily. Each cycle is 28 days.
Period: Overall Study
Arm/Group | Erlotinib + BKM120
Started | 37
Completed | 0
Not Completed | 37
Not completed — Adverse Event | 8
Not completed — Withdrawal by Subject | 5
Not completed — Disease Progression | 21
Not completed — Death | 2
Not completed — Still on Treatment | 1

BASELINE CHARACTERISTICS:
Population: Patients that have received at least one dose of study treatment
Arm/Group | Erlotinib + BKM120
Number analyzed (Participants) | 37
Age, Continuous [Median (Full Range); unit: years] | 69 [42 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37
Smoking Status [Count of Participants; unit: Participants]
  Never smoker | 19
  Current smoker | 2
  Former smoker | 16

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival at 3 Months
Description: Percentage of patients who are alive and progression-free at 3 months (APF3) from first treatment.
Time Frame: 3 months
Population: Patients that were treated with at least one dose of study treatment
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib + BKM120
Number analyzed (Participants) | 37
percentage of participants | 50.4

2. Secondary Outcome: Overall Survival
Description: Defined as the time from first treatment until death from any cause.
Time Frame: every 3 months after study treatment, projected 24 months
Population: Patients that received at least one dose of study treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib + BKM120
Number analyzed (Participants) | 37
months | 12.2 [7.2 to 33.3]

3. Secondary Outcome: Duration of Response
Description: Defined as the time from complete or partial response (CR or PR) until objective tumor progression. Tumor measurements will be obtained using CT scans of chest, abdomen and pelvis and assessed per RECIST v 1.1. Complete response (CR) is defined as a disappearance of all lesions; partial response (PR) is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking the baseline sum LD as reference. Stable Disease (SD) is defined as neither sufficient shrinkage to qualify for PR, nor sufficient increase to qualify for progressive disease, taking as reference the smallest (nadir) sum LD since start of treatment.
Time Frame: every 8 weeks for 12 months, then every 12 weeks thereafter, estimated 18 months
Population: Of 37 participates that received study treatment, only two participants met the minimum criteria to be included (one censored, and the remaining one analyzed for duration of response)
Measure: Number; unit: months
Arm/Group | Erlotinib + BKM120
Number analyzed (Participants) | 1
months | 3.2

4. Secondary Outcome: Objective Response Rate
Description: Defined as the percentage of complete and partial responses (CR + PR) among all patients. Complete response (CR) is defined as a disappearance of all lesions; partial response (PR) is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking the baseline sum LD as reference. Stable Disease (SD) is defined as neither sufficient shrinkage to qualify for PR, nor sufficient increase to qualify for progressive disease, taking as reference the smallest (nadir) sum LD since start of treatment.
Time Frame: every 8 weeks for 12 months, then every 12 weeks thereafter, estimated 18 months
Population: patients that received at least one dose of study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Erlotinib + BKM120
Number analyzed (Participants) | 37
percentage of participants | 5.4 [0.7 to 18.2]

5. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events as a Measure of Safety.
Description: Adverse events will be graded using CTCAE v4.3. and will be collected until 30 days after the discontinuation of study treatment for each participant. A non-serious adverse event is any untoward medical occurrence. A serious adverse event (SAE) is an event that meets one or more of the following: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; requires intervention to prevent permanent impairment or damage. Specific AE and SAE terms are provided in the Adverse event module.
Time Frame: Every 2 weeks for 8 weeks, then every 8 weeks thereafter, estimated 24 months
Population: Patients that received at least one dose of study treatment
Measure: Number; unit: participants
Arm/Group | Erlotinib + BKM120
Number analyzed (Participants) | 37
participants
  Adverse Events (all grades) | 37
  Serious Adverse Events | 13

ADVERSE EVENTS:
Time Frame: Collected from the date of first treatment until 30 days after the discontinuation of study treatment, approximately months
Arm/Group | Erlotinib + BKM120
Serious Adverse Events (participants affected / at risk) | 13/37
Other Adverse Events (participants affected / at risk) | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erlotinib + BKM120 (N=37)
Asthenia (General disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Disease progression (General disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Pyrexia (General disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Vasogenic cerebral oedema (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib + BKM120 (N=37)
Diarrhoea (Gastrointestinal disorders) | 29
Fatigue (General disorders) | 20
Nausea (Gastrointestinal disorders) | 17
Decreased Appetite (Metabolism and nutrition disorders) | 14
Rash (Skin and subcutaneous tissue disorders) | 10
Dehydration (Metabolism and nutrition disorders) | 9
Hyperglycaemia (Metabolism and nutrition disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dysgeusia (Nervous system disorders) | 8
Dyspepsia (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 7
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Dry Skin (Skin and subcutaneous tissue disorders) | 6
Headache (Nervous system disorders) | 6
Weight Decreased (Investigations) | 6
Hypokalaemia (Metabolism and nutrition disorders) | 5
Oedema Peripheral (General disorders) | 5
Dizziness (Nervous system disorders) | 5
Depression (Psychiatric disorders) | 5
Insomnia (Psychiatric disorders) | 5
Abdominal Pain (Gastrointestinal disorders) | 4
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 4
Asthenia (General disorders) | 4
Anxiety (Psychiatric disorders) | 4
Pneumonia (Infections and infestations) | 4
Urinary Tract Infection (Infections and infestations) | 4
Constipation (Gastrointestinal disorders) | 3
Dry Mouth (Gastrointestinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 3
Mucosal Inflammation (General disorders) | 3
Pain (General disorders) | 3
Pyrexia (General disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3
Confusional State (Psychiatric disorders) | 3
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3
Alanine Aminotransferase Increased (Investigations) | 3
Deep Vein Thrombosis (Vascular disorders) | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2
Chest Pain (General disorders) | 2
Nail Disorder (Skin and subcutaneous tissue disorders) | 2
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 2
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 2
Lower Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2
Syncope (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 2
Irritability (Psychiatric disorders) | 2
Mood Altered (Psychiatric disorders) | 2
Upper Respiratory Tract Infection (Infections and infestations) | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2
Dysuria (Renal and urinary disorders) | 2
Pollakiuria (Renal and urinary disorders) | 2
Supraventricular Tachycardia (Cardiac disorders) | 2
Eye Pain (Eye disorders) | 2
Vision Blurred (Eye disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.